CLINICAL TRIAL: NCT03200041
Title: Clinical Evaluation of the IONA Test for Non-invasive Pre Natal Screening in Twin Pregnancies
Acronym: TWIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Premaitha Health (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: PMH/0915/01
Record Dates: First submitted 2016-04-25; First posted 2017-06-27 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Down Syndrome; Patau Syndrome; Edward's Syndrome
MeSH Terms: conditions — Down Syndrome; Trisomy 13 Syndrome; Trisomy 18 Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Risk (Other): 350 Low risk The only intervention is a 20 ml blood sample will be taken from each participant.
  Interventions: Procedure: Blood sample
- High Risk (Other): 150 High Risk going onto invasive diagnostic procedure. The only intervention is a 20 ml blood sample will be taken from each participant.
  Interventions: Procedure: Blood sample

INTERVENTIONS:
Procedure: Blood sample — 20 ml blood sample taken from vein in arm

SUMMARY:
The purpose of this study is to evaluate the performance of the IONA® test which is a non-invasive prenatal test (NIPT) for Down's syndrome and other chromosomal abnormalities in twin pregnancies, from a maternal blood sample.

DETAILED DESCRIPTION:
350 low risk and 150 high risk women with twin pregnancies will be recruited to produce a large cohort evaluation the use of the IONA test in twin pregnancies for Downs, Edwards and Patau syndrome. Reserve samples will also be used to further develop the test for other chromosomal abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* Currently pregnant with twin foetuses at time of entry to study
* Have had or are about to have a conventional screening test (combined/quad test, ultrasound scan or other NIPT)
* If identified as high risk, intend to undergo prenatal invasive diagnosis and/or undergoing invasive prenatal therapy such as laser treatment for TTTS where a sample of amniotic fluid is taken for karyotyping.

Exclusion Criteria:

* Participant herself has down syndrome or other chromosomal abnormality

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2016-02; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Number of IONA test results which are concordant or discordant with Invasive test or Birth outcome. | 18 months
  IONA test results will be compared to Karyotyping from birth outcome and invasive procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Asma Khalil, MBBS, Principal Investigator — National Health Service, United Kingdom
Locations (1):
- Premaitha Health, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IONA Test results being given to patients